CLINICAL TRIAL: NCT00061893
Title: A Pilot Study of Low-Dose Antiangiogenic Chemotherapy in Combination With Standard Multiagent Chemotherapy for Patients With Newly Diagnosed Metastatic Ewing Sarcoma Family of Tumors
Brief Title: Vinblastine, Celecoxib, and Combination Chemotherapy in Treating Patients With Newly-Diagnosed Metastatic Ewing's Sarcoma Family of Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEWS02P1; CDR0000302409 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Sarcoma
Keywords: metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Celecoxib; Cyclophosphamide; Doxorubicin; Etoposide; Ifosfamide; Vinblastine; Vincristine; Radiotherapy; Mesna; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination chemotherapy (Experimental): Metastatic Ewing Sarcoma - 14-cycle study building on conventional tx (cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, ifosfamide, etoposide) and adding two antiangiogenic agents: the vinca alkaloid vinblastine and the cyclooxygenase-2 inhibitor celecoxib. Refer to the Interventions section for dosages, method of delivery and frequency of administration.
  Interventions: Drug: celecoxib; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: vinblastine sulfate; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: radiation therapy; Drug: MESNA; Drug: Filgrastim

INTERVENTIONS:
Drug: celecoxib — Given orally, Celecoxib 250 mg/m2 PO BID (500mg/m2/day) from Day 1 of Cycle 1 through Day 21 of Cycle 14. The dose should be rounded off to the nearest 100 mg. If PK studies are being done, Celecoxib should be given 24 hours prior to the other drugs for Cycle 1 only. [Celecoxib may be interrupted for up to 7 days around the time of surgical procedures.] .
Drug: cyclophosphamide — Given IV, 1200 mg/m2 IV infusion over 1 hour with MESNA uroprotection, on Day 1. For children < 1 year treat with 50% doses calculated on a m2 basis. If tolerated (no delay in administration of the next cycle due to delayed count recovery or delayed resolution of other toxicities and no serious toxicities), consider increasing to 75% and then to 100% of the calculated full dose.
Drug: doxorubicin hydrochloride — Given IV, Doxorubicin 75 mg/ m2 /course continuous IV infusion over 48 hours, beginning Day 1. Note: The total doxorubicin dose per cycle is 75 mg/ m2, which will be given as 37.5 mg/m2/day x 2 days. Doxorubicin may be given as a continuous infusion or brief infusion.
Drug: etoposide — Given IV, Vincristine 2 mg/m2 IV push, on Day 1. Maximum dose 2 mg. For children < 1 year treat with 50% doses calculated on a m2 basis. If tolerated (no delay in administration of the next cycle due to delayed count recovery or delayed resolution of other toxicities and no serious toxicities), consider increasing to 75% and then to 100% of the calculated full dose.
Drug: ifosfamide — Given IV,Ifosfamide 1800 mg/m2 /day IV infusion over 1 hour, Days 1-5 of each cycle. (9,000 mg/m2 max total dose per cycle). Prehydrate for 6 hours, 1,000 ml/m2 total volume (165 ml/m2/hour for 6 hours). For children < 1 year treat with 50% doses calculated on a m2 basis. If tolerated (no delay in administration of the next cycle due to delayed count recovery or delayed resolution of other toxicities and no serious toxicities), consider increasing to 75% and then to 100% of the calculated full dose.
Drug: vinblastine sulfate — Given IV, Vinblastine 1 mg/m2/d IV push three times per week beginning Day 1 of Cycle 1 and continuing through Day 21 of Cycle 14. In weeks during which vincristine is given, hold one dose of vinblastine and administer only 2 doses of vinblastine during that week. If vinblastine is due the same day as vincristine, hold that dose of vinblastine. [Vinblastine may be interrupted for up to 7 days around the time of surgical procedures.]
Drug: vincristine sulfate — Given IV, Vincristine 2 mg/m2 IV push, on Day 1. Maximum dose 2 mg. For children < 1 year treat with 50% doses calculated on a m2 basis. If tolerated (no delay in administration of the next cycle due to delayed count recovery or delayed resolution of other toxicities and no serious toxicities), consider increasing to 75% and then to 100% of the calculated full dose.
Procedure: conventional surgery — Patients who respond to induction chemotherapy undergo surgery on week 13. Patients who have inadequate margins after surgery undergo radiotherapy beginning on week 15. (see Detailed Description for frequency of administration and groups evaluated)
Radiation: radiation therapy — Patients with unresectable lesions undergo radiotherapy 5 days a week for approximately 6 weeks beginning on week 13. (see Detailed Description for frequency of administration and groups evaluated)
Drug: MESNA — The total daily MESNA dose is equal to at least 60% of the daily cyclophosphamide or ifosfamide dose, or by continuous infusion of the 60% dose. MESNA continuous infusion should be started at the same time as the cyclophosphamide/ifosfamide and be completed no sooner than 8 hours after the end of the cyclophosphamide or ifosfamide infusion. The oral dose of MESNA is 2x the IV dose. Patients able to tolerate oral MESNA may receive the final dose by mouth at 40% of the oxazaphosphorine (cyclophosphamide or ifosfamide) dose. The dose should be given two hours earlier than the IV dose would be given. Additionally, if the patient vomits within two hours after the oral dose, the dose should be repeated or IV MESNA given.
Drug: Filgrastim — G-CSF (Filgrastim) 5 micrograms/kg/day subcutaneously beginning 24 to 48 hours after the last dose of chemotherapy, and continuing until the absolute neutrophil count is 2,000/µL or greater after nadir.
  Other Names: G-CSF

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinblastine, work in different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may stop the growth of Ewing's sarcoma by stopping blood flow to the tumor. Combining more than one chemotherapy drug with celecoxib may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining low-dose vinblastine and celecoxib with standard regimens of combination chemotherapy in treating patients who have newly-diagnosed metastatic Ewing's sarcoma family of tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and safety of low-dose vinblastine and celecoxib in combination with standard multiagent chemotherapy in patients with newly diagnosed metastatic Ewing's sarcoma family of tumors.
* Determine the event-free survival of patients treated with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a pilot, multicenter study.

* Induction therapy: Patients receive the following alternating regimens:

  * VAC (courses 1 and 3): Patients receive vincristine IV and cyclophosphamide IV over 1 hour on day 1 and doxorubicin IV continuously on days 1 and 2 of weeks 1 and 7.
  * IE (courses 2 and 4): Patients receive ifosfamide IV over 1 hour and etoposide IV over 1-2 hours on days 1-5 of weeks 4 and 10.

Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning 24-48 hours after the last dose of chemotherapy and continuing until blood counts recover.

Treatment repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity.

* Local control and consolidation therapy: Beginning on week 13, patients are assigned to 1 of 4 regimens based on disease status.

  * Regimen A (surgery only): Patients who respond to induction chemotherapy undergo surgery on week 13. Patients then begin consolidation therapy on week 15 with the following alternating regimens:

    * VAC (courses 5, 7, and 9): Patients receive VAC on weeks 15, 21, and 27.
    * IE (courses 6, 8, 10, 12, and 14): Patients receive IE on weeks 18, 24, 30, 36, and 42.
    * VC (courses 11 and 13): Patients receive vincristine IV and cyclophosphamide IV over 1 hour on weeks 33 and 39.
  * Regimen B (radiotherapy only): Patients with unresectable lesions undergo radiotherapy once daily 5 days a week for up to approximately 6 weeks beginning on week 13. Patients also receive consolidation therapy beginning on week 13, with the following alternating regimens:

    * VAC (courses 5, 9, and 11): Patients receive VAC on weeks 13, 25, and 31.
    * IE (courses 6, 8, 10, 12, and 14): Patients receive IE on weeks 16, 22, 28, 34, and 40.
    * VC (courses 7 and 13): Patients receive VC on weeks 19 and 37.
  * Regimen C (surgery and radiotherapy): Patients who respond to induction chemotherapy undergo surgery on week 13. Patients who have inadequate margins after surgery undergo radiotherapy (as in regimen B) beginning on week 15. Patients also receive consolidation therapy, beginning on week 15, with the following alternating regimens:

    * VAC (courses 5, 9, and 11): Patients receive VAC on weeks 15, 27, and 33.
    * IE (courses 6, 8, 10, 12, and 14): Patients receive IE on weeks 18, 24, 30, 36, and 42.
    * VC (courses 7 and 13): Patients receive VC on weeks 21 and 39.
  * Regimen D (preoperative radiotherapy): Patients with bulky lesions who do not have a good clinical and radiographic response to induction therapy begin consolidation therapy on week 13 with VAC (course 5) and undergo concurrent radiotherapy as in regimen B. Patients then receive IE on weeks 16 and 19 for courses 6 and 7. Patients undergo surgery on week 22. Patients continue consolidation therapy with the following alternating regimens:

    * VAC (courses 8 and 9): Patients receive VAC on weeks 24 and 27.
    * IE (courses 10, 12, and 14): Patients receive IE on weeks 30, 36, and 42.
    * VC (courses 11 and 13): Patients receive VC on weeks 33 and 39. Patients receive G-CSF SC (as in induction therapy) during all consolidation courses.

Consolidation therapy continues for 10 courses in the absence of disease progression or unacceptable toxicity.

* Vinblastine and celecoxib therapy: Throughout induction, local control, and consolidation therapies, patients also receive vinblastine IV 3 times a week (twice a week during the weeks that vincristine is given) and oral celecoxib twice daily, beginning on day 1 of course 1 and continuing until the completion of course 14.* NOTE: *To assess for safety, the first 6 patients enrolled receive vinblastine only during courses 1 and 2 and celecoxib is then added for all subsequent courses.

Patients are followed every 3 months for 3 years and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 6-36 patients will be accrued for this study within 1.17 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed Ewing's sarcoma family of tumors of the bone or soft tissues

  * Paraspinal tumors of extra-dural origin and Askin's tumor of the chest wall are eligible
* Metastatic disease, defined by the following criteria:

  * Lesions are discontinuous from the primary tumor, are not regional lymph nodes, and do not share a body cavity with the primary tumor
  * A single pulmonary or pleural nodule greater than 1 cm OR multiple nodules greater than 0.5 cm are considered evidence of pulmonary or pleural metastases (unless there is another clear medical explanation for these lesions)
  * Contralateral pleural effusions are considered metastatic disease
* No CNS involvement

PATIENT CHARACTERISTICS:

Age

* 50 and under (at diagnosis)

Performance status

* Lansky 50-100% (under 17 years of age)
* Karnofsky 50-100% (age 17 and over)

  * Patients whose performance status is affected by a pathological fracture are allowed provided they are able to undergo treatment

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT less than 5 times ULN

Renal

* Creatinine adjusted according to age as follows*:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months -11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male]) OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min* NOTE: *Unless these values are related to renal insufficiency secondary to tumor involvement that is expected to improve once the tumor mass is smaller (e.g., pelvic mass causing obstructive hydronephrosis)

Cardiovascular

* Shortening fraction at least 27% by echocardiogram OR
* Ejection fraction at least 50% by MUGA

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Body surface area at least 0.4 m^2
* No allergy to sulfa
* No aspirin hypersensitivity
* No asthma triad (asthma with nasal polyps, and urticaria)
* No other prior cancer, including nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior bone marrow or stem cell transplantation

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Other

* No other concurrent nonsteroidal anti-inflammatory medications, including salicylates
* No concurrent dexrazoxane unless approved by the study investigator

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2004-04; Primary Completion 2008-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy L. Felgenhauer, MD, PS, Study Chair — Sacred Heart Children's Hospital
Locations (101):
- United States (87):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - University of California Davis Cancer Center, Sacramento, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - OU Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales, Australia
- Canada (12):
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Result] Felgenhauer JL, Nieder ML, Krailo MD, Bernstein ML, Henry DW, Malkin D, Baruchel S, Chuba PJ, Sailer SL, Brown K, Ranganathan S, Marina N. A pilot study of low-dose anti-angiogenic chemotherapy in combination with standard multiagent chemotherapy for patients with newly diagnosed metastatic Ewing sarcoma family of tumors: A Children's Oncology Group (COG) Phase II study NCT00061893. Pediatr Blood Cancer. 2013 Mar;60(3):409-14. doi: 10.1002/pbc.24328. Epub 2012 Oct 12. PMID 23065953

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Chemotherapy: Metastatic Ewing Sarcoma - 14-cycle study building on conventional tx (cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, ifosfamide, etoposide) and adding two antiangiogenic agents: the vinca alkaloid vinblastine and the cyclooxygenase-2 inhibitor celecoxib. Angiogenesis may be a suitable target for cancer therapy because tumor growth is partially dependent upon neovascularization. Vinblastine sulfate has been shown to have antiangiogenic activity and in preclinical studies, celecoxib has demonstrated antiangiogenic activity as well as inducing apoptosis in tumor vessel endothelial cells. The feasibility and safety of adding antiangiogenic agents to conventional chemotherapy will be assessed by imaging studies (DeMRI, PET, Thallium scintigraphy). Local control with conventional surgery, radiation therapy or both will be tailored for each patient to optimally treat all sites of disease.
Period: Overall Study
Arm/Group | Combination Chemotherapy
Started | 38
Completed | 20
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Combination Chemotherapy
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.97 (5.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 34
  Canada | 4

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Severe Toxicity
Description: An incidence of severe toxicity is defined to be the occurrence of grade 3 or higher infection or grade 3 or higher sensory neuropathy during cycles 1-2 of protocol therapy. If 12 or more patients experience grade 3 or higher infection or five or more patients experience grade 3 or higher sensory neuropathy during cycles 1-2 of protocol therapy, the regimen will be flagged as being associated with an excessive rate of severe toxicity.
Time Frame: The first two cycles (6 weeks) of protocol chemotherapy
Population: By protocol design, all eligible patients who received protocol therapy were considered in the evaluation of severe toxicity. Three (3) patients were considered ineligible. All other patients (35) started protocol therapy and are thus included in the evaluation for this measure.
Measure: Number; unit: participants
Arm/Group | Combination Chemotherapy
Number analyzed (Participants) | 35
participants
  Grade 3 or Higher Infection | 1
  Grade 3 or Higher Sensory Neuropathy | 1

2. Secondary Outcome: Event Free Survival
Time Frame: 24 months after start of protocol therapy
Population: By protocol design, all eligible patients who received protocol therapy were considered in the evaluation of Event Free Survival. Three (3) patients were considered ineligible. All other patients (35) started protocol therapy and are thus included in the evaluation for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination Chemotherapy
Number analyzed (Participants) | 35
percentage of participants | 35 [19 to 51]

ADVERSE EVENTS:
Description: By protocol design, all eligible patients who received any protocol therapy were considered in the evaluation of study outcome measures, including the occurence of Adverse Events. Three (3) patients were considered ineligible. The remaining eligible 35 patients started protocol therapy and are included in the valuation of Adverse Event experience.
Arm/Group | Combination Chemotherapy
Serious Adverse Events (participants affected / at risk) | 33/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Chemotherapy (N=35)
Abdominal pain (Gastrointestinal disorders) | 2 — Grades 3-5
Activated partial thromboplastin time prolonged (Investigations) | 1 — Grades 3-5
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 — Grades 3-5
Alanine aminotransferase increased (Investigations) | 2 — Grades 3-5
Anemia (Blood and lymphatic system disorders) | 12 — Grades 3-5
Anorexia (Metabolism and nutrition disorders) | 6 — Grades 3-5
Aspartate aminotransferase increased (Investigations) | 2 — Grades 3-5
Back pain (Musculoskeletal and connective tissue disorders) | 1 — Grades 3-5
Bladder infection (Infections and infestations) | 1 — Grades 3-5
Bladder spasm (Renal and urinary disorders) | 1 — Grades 3-5
Blood bilirubin increased (Investigations) | 3 — Grades 3-5
Bronchial infection (Infections and infestations) | 1 — Grades 3-5
Catheter related infection (Infections and infestations) | 2 — Grades 3-5
Colitis (Gastrointestinal disorders) | 1 — Grades 3-5
Constipation (Gastrointestinal disorders) | 2 — Grades 3-5
Cystitis noninfective (Renal and urinary disorders) | 1 — Grades 3-5
Dehydration (Metabolism and nutrition disorders) | 4 — Grades 3-5
Diarrhea (Gastrointestinal disorders) | 4 — Grades 3-5
Dysphagia (Gastrointestinal disorders) | 3 — Grades 3-5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 — Grades 3-5
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 — Grades 3-5
Esophagitis (Gastrointestinal disorders) | 2 — Grades 3-5
Fatigue (General disorders) | 1 — Grades 3-5
Febrile neutropenia (Blood and lymphatic system disorders) | 15 — Grades 3-5
Fever (General disorders) | 1 — Grades 3-5
Fibrinogen decreased (Investigations) | 1 — Grades 3-5
Forced expiratory volume decreased (Investigations) | 1 — Grades 3-5
Gastritis (Gastrointestinal disorders) | 3 — Grades 3-5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — Grades 3-5
GGT increased (Investigations) | 2 — Grades 3-5
Hematuria (Renal and urinary disorders) | 3 — Grades 3-5
Hyperglycemia (Metabolism and nutrition disorders) | 1 — Grades 3-5
Hyperkalemia (Metabolism and nutrition disorders) | 1 — Grades 3-5
Hypermagnesemia (Metabolism and nutrition disorders) | 1 — Grades 3-5
Hypernatremia (Metabolism and nutrition disorders) | 1 — Grades 3-5
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 — Grades 3-5
Hypocalcemia (Metabolism and nutrition disorders) | 2 — Grades 3-5
Hypokalemia (Metabolism and nutrition disorders) | 14 — Grades 3-5
Hypomagnesemia (Metabolism and nutrition disorders) | 1 — Grades 3-5
Hyponatremia (Metabolism and nutrition disorders) | 6 — Grades 3-5
Hypophosphatemia (Metabolism and nutrition disorders) | 3 — Grades 3-5
Hypotension (Vascular disorders) | 3 — Grades 3-5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 — Grades 3-5
Ileus (Gastrointestinal disorders) | 1 — Grades 3-5
Infections and infestations - Other, specify (Infections and infestations) | 18 — Grades 3-5
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 — Grades 3-5
Lung infection (Infections and infestations) | 1 — Grades 3-5
Lymphocyte count decreased (Investigations) | 2 — Grades 3-5
Mucositis oral (Gastrointestinal disorders) | 3 — Grades 3-5
Myocardial infarction (Cardiac disorders) | 1 — Grades 3-5
Nausea (Gastrointestinal disorders) | 3 — Grades 3-5
Neutrophil count decreased (Investigations) | 19 — Grades 3-5
Pain of skin (Skin and subcutaneous tissue disorders) | 1 — Grades 3-5
Pericardial effusion (Cardiac disorders) | 1 — Grades 3-5
Perineal pain (Reproductive system and breast disorders) | 1 — Grades 3-5
Peripheral motor neuropathy (Nervous system disorders) | 1 — Grades 3-5
Peripheral sensory neuropathy (Nervous system disorders) | 2 — Grades 3-5
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 — Grades 3-5
Platelet count decreased (Investigations) | 16 — Grades 3-5
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 — Grades 3-5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 — Grades 3-5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 — Grades 3-5
Sepsis (Infections and infestations) | 1 — Grades 3-5
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 — Grades 3-5
Upper respiratory infection (Infections and infestations) | 1 — Grades 3-5
Urinary retention (Renal and urinary disorders) | 1 — Grades 3-5
Urinary tract infection (Infections and infestations) | 2 — Grades 3-5
Vascular access complication (Injury, poisoning and procedural complications) | 1 — Grades 3-5
Vasovagal reaction (Nervous system disorders) | 1 — Grades 3-5
Vomiting (Gastrointestinal disorders) | 4 — Grades 3-5
Weight loss (Investigations) | 4 — Grades 3-5
White blood cell decreased (Investigations) | 16 — Grades 3-5
Wound infection (Infections and infestations) | 1 — Grades 3-5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Chemotherapy (N=35)
Acidosis (Metabolism and nutrition disorders) | 9 — Grades 1-2
Activated partial thromboplastin time prolonged (Investigations) | 1 — Grades 1-2
Alanine aminotransferase increased (Investigations) | 3 — Grades 1-2
Anemia (Blood and lymphatic system disorders) | 2 — Grades 1-2
Aspartate aminotransferase increased (Investigations) | 1 — Grades 1-2
Bladder spasm (Renal and urinary disorders) | 1 — Grades 1-2
Blood bilirubin increased (Investigations) | 2 — Grades 1-2
Burn (Injury, poisoning and procedural complications) | 1 — Grades 1-2
Catheter related infection (Infections and infestations) | 1 — Grades 1-2
Constipation (Gastrointestinal disorders) | 1 — Grades 1-2
Depression (Psychiatric disorders) | 1 — Grades 1-2
Gastritis (Gastrointestinal disorders) | 8 — Grades 1-2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 — Grades 1-2
Hematuria (Renal and urinary disorders) | 12 — Grades 1-2
Hyperglycemia (Metabolism and nutrition disorders) | 2 — Grades 1-2
Hypermagnesemia (Metabolism and nutrition disorders) | 1 — Grades 1-2
Hypertension (Vascular disorders) | 1 — Grades 1-2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 — Grades 1-2
Hypocalcemia (Metabolism and nutrition disorders) | 3 — Grades 1-2
Hypokalemia (Metabolism and nutrition disorders) | 9 — Grades 1-2
Hypophosphatemia (Metabolism and nutrition disorders) | 17 — Grades 1-2
Infections and infestations - Other, specify (Infections and infestations) | 1 — Grades 1-2
INR increased (Investigations) | 1 — Grades 1-2
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 2 — Grades 1-2
Mucositis oral (Gastrointestinal disorders) | 1 — Grades 1-2
Peripheral motor neuropathy (Nervous system disorders) | 2 — Grades 1-2
Peripheral sensory neuropathy (Nervous system disorders) | 4 — Grades 1-2
Proctitis (Gastrointestinal disorders) | 1 — Grades 1-2
Proteinuria (Renal and urinary disorders) | 15 — Grades 1-2
Psychosis (Psychiatric disorders) | 1 — Grades 1-2
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 — Grades 1-2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 — Grades 1-2
Thromboembolic event (Vascular disorders) | 1 — Grades 1-2
Urinary frequency (Renal and urinary disorders) | 1 — Grades 1-2
Urinary tract infection (Infections and infestations) | 1 — Grades 1-2
Urinary tract pain (Renal and urinary disorders) | 1 — Grades 1-2
Vomiting (Gastrointestinal disorders) | 2 — Grades 1-2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No